CLINICAL TRIAL: NCT01939392
Title: Rapid Renal Sympathetic Denervation for Resistant Hypertension Using the OneShot Renal Denervation System II
Brief Title: Rapid Renal Sympathetic Denervation for Resistant Hypertension II
Acronym: RAPID II
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-1003
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Resistant Hypertension; Uncontrolled Hypertension; Renal Artery Ablation
Keywords: Resistant hypertension; Uncontrolled hypertension; Renal artery ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal Denervation (Experimental): Subjects randomized to the Renal Denervation arm will receive bilateral renal ablation with the OneShot system and be maintained on antihypertensive medication.
  Interventions: Device: Renal Denervation (OneShot™ Renal Denervation System)
- Optimal Medical Therapy (No Intervention): Subjects randomized to the control arm will be maintained on antihypertensive medications.

INTERVENTIONS:
Device: Renal Denervation (OneShot™ Renal Denervation System)
  Other Names: OneShot Ablation system; Catheter-based renal denervation
  Arms: Renal Denervation

SUMMARY:
This is a global, multi-center, prospective, randomized, controlled study of the safety and effectiveness of renal denervation with the OneShot Renal Denervation System in patients with uncontrolled hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Individual has a systolic blood pressure ≥ 160 mmHg based on an average of three office blood pressure readings.
* Stable drug regimen including three or more anti-hypertensive medications including a diuretic

Exclusion Criteria:

* Renal anatomy unsuitable for treatment
* Presence of hemodynamically significant valvular heart disease for which reduction of blood pressure would be considered hazardous
* Patient has Type I diabetes
* Has scheduled or planned surgery within the next 6 months
* Individual is pregnant nursing or plans to be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Major adverse event (MAE) rate through 30 days post randomization | 30 days
Change in office systolic blood pressure (SBP) from baseline to 6 months post-randomization | 6 months

SECONDARY OUTCOMES:
Acute Procedural Safety | 30 days
Chronic procedural safety | 6 months
Reduction in SBP by >10 mmHg at 6 months | 6 months
Changes in office SBP and diastolic blood pressure (DBP) from baseline to follow-up visits | 6, 12, 24, and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, MD, Principal Investigator — Park-Krankenhaus Liepzig; Guiseppe Mancia, MD, Principal Investigator — Universita Minano-Bicocca, Ospedale San Gerardo di Monza
Locations (1):
- Hospital San Raffaele, Milan, Italy